CLINICAL TRIAL: NCT02364492
Title: An Open Label First-in-Human Adjuvant Phase I Study of a Synthetic Multiple Antigenic Glycopeptide Displaying a Tri Tn Glycotop (MAG-Tn3) Plus AS15, as a Therapeutic Vaccine Candidate in Patients With Non Metastatic, HER2 Negative Localized Breast Cancer at High-Risk of Relapse
Brief Title: A Phase I Study of a Therapeutic Vaccine Candidate in Patients With Localized Breast Cancer at High-Risk of Relapse
Acronym: MAGTRIVACSEIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.14
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2021-07

CONDITIONS: Breast Neoplasms
Keywords: [C04.588.180]
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MAG-Tn3 + AS15 (Experimental): 3 escalating doses of MAG-Tn3 in combination with a fixed dose of AS15 adjuvant.
  For each dose patient will receive 6 injections at 3 interval weeks.
  Interventions: Drug: MAG-TN3 + AS15

INTERVENTIONS:
Drug: MAG-TN3 + AS15

SUMMARY:
The purpose of this study is to evaluate if a maximum tolerated dose (MTD) can be obtained following 2 administrations of the MAG-Tn3 + AS15 cancer vaccine when administered at doses of 30 µg, 100 µg or 300 µg IM every three weeks.

DETAILED DESCRIPTION:
This study is a three dose level open-label, non-randomized, dose-escalation study Phase I of the safety of the vaccine candidate MAG-Tn3 + AS15 administered to patients with HER2 negative, high-risk localized breast cancer in remission.

A maximum of 30 patients will be included in the study:

* 3 or 6 patients in the 1st dose level (30 µg)
* 6 or 12 patients in the 2nd dose level (100 µg)
* 6 or 12 patients in the 3rd dose level (300 µg) The clinical study phase I is composed of a vaccination period of about 4 months (16 weeks) and a follow-up period of 36 months (3 years).

Each patient will receive one of the three escalating doses of MAG-Tn3 in combination with a fixed dose of AS15 adjuvant.

The subject will receive 6 vaccine injections, administered by intramuscular injection with a 3-weeks interval between injections. Each patient will be followed 36 months after the last injection. The follow-up period is composed of a short-term follow-up period of 6 months and a long-term follow-up period of 30 months.

A total of 20 visits will be required for each patient. Clinical data and blood samples will be collected for analysis for each patient.

Clinical study data will be recorded for each patient on source documentation and then entered on electronic CRFs (eCRFs) using a proprietary Electronic Data Capture (EDC) Clinical Data Base Software System. The eCRF data are to be entered by site personnel trained in EDC data entry.

A monitor will visit the site regularly to check the completeness of patient records, the accuracy of entries on the e-CRFs, the adherence to the protocol and to Good Clinical Practice, the progress of enrollment, and to ensure that study drug is being stored, dispensed, and accounted for according to specifications.

Institut Pasteur or designated CRO will conduct data management. Data entered into EDC will be housed in a central database. Changes will be tracked to provide an audit trail. Interactive data checks will be carried out as applicable during the data entry process. Additional data checks are programmed to identify errors in the SAS datasets. Applicable queries based on the SAS datasets will be added to EDC for resolution by data management personnel. At the conclusion of the study, when all data have been entered and source document verified, with no outstanding queries remaining, the Investigator of each site will be required to electronically sign each patient's casebook to confirm that the data for each patient are complete and accurate and consistent with the patient's source documents. The data will then be locked to prevent further editing.

Concomitant medications entered into the database will be coded using the WHO Drug Reference List, which employs the Anatomical Therapeutic Chemical classification system. Medical history/current medical conditions and adverse events terminology will be coded using the Medical dictionary for regulatory activities.The newest version of the dictionary at data base lock will be used.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a diagnosis of epithelial breast carcinoma which is, according to TNM classification:

   * Any T
   * With Positive (N+) or Negative (N-) Lymph-Node depending on the patient profile (see below criteria n°3)
   * And Non metastatic (M0)
2. HER2/neu-negative (Immunohistochemical expression "0-1+", and/or FISH/CISH "non amplified" according to ASCO 2012 criteria)
3. First line treatment population with a High-Risk of Relapse as defined by:

   * with at least one positive lymph nodes (LN) at primary surgery
   * or after completion of 6-8 cycles of anthracyclins/taxanes-based neoadjuvant chemotherapy

   OR

   Negative hormone receptors: ER- and PR- , (<10%), i.e "Triple Negative breast cancer"
4. Patients must have completed all their local and regional treatments including adequate surgery and radiation therapy, and at least 6 cycles of chemotherapy (neoadjuvant and/or adjuvant) according to institutional and national standards.
5. The time interval between the end of all the first line standard treatment (completion of surgery, chemotherapy and radiation therapy) should be at least 1 month and within a maximum of 18 months before inclusion in the study.
6. Patients eligible to adjuvant hormone therapy should have started their treatment for at least 2 months at the time of inclusion in the study.
7. Patients treated by biphosphonates should have started their treatment for at least 28 days at the time of inclusion in the study
8. Patients must be free of any breast cancer recurrence as shown by standard diagnostic tests at the entry into the study.
9. Patients should have an expected life expectancy of at least 12 months as evaluated by the investigator at the entry into the study.
10. Written informed consent must be obtained prior to any protocol-specific procedures.
11. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
12. Patients must not be pregnant. Non-menopausal women must have a negative pregnancy test prior to enrolment, and must use adequate contraception (1 barrier method) throughout the study.
13. Patients must be aware of the potential harm of the study treatment on any future pregnancy and must agree not to become pregnant within 24 months following the last study vaccine injection.
14. Patients must not be lactating.
15. Patients must be between 18 and 70 years of age.
16. Patients must have adequate bone marrow reserve (testing within 2 weeks before inclusion) as evaluated by the investigator.

    WBC ≥3000/mm3, neutrophils ≥1500/mm3, platelets ≥100,000/mm3, and hemoglobin ≥10 g/dL.
17. Patients must have an absolute lymphocytes count >800 cells/mm3
18. Patients with creatinine clearance considerate as normal as evaluated by the investigator calculated creatinine clearance > 50 ml/min (using the Cockcroft-Gault Formula)
19. Patients must have adequate hepatic function as evaluated by the investigator serum total bilirubin <1.5* times the upper limit of normal (ULN), AST and ALT < 3* times the ULN, and alkaline phosphatases<2.5* times, the ULN. Patients with an alkaline phosphatase above normal must have negative bone scans and abdominal CT scans prior to entry onto the study.

    * biological limit values specified into the NCI-CTCAE V4.03 of June 2010
20. Before inclusion patients must have negative test for HIV1 and HIV2; no history of active hepatitis B or C and no chronic hepatitis B or C requiring treatment with antiviral therapy
21. The patients must be covered by national social security insurance.
22. In the view of the investigator, the patients can and will comply with the requirements of this protocol.

Exclusion Criteria:

1. Any breast cancer recurrence or metastasis.
2. Patients with HER2/neu positive breast carcinoma (IHC score 2+ or 3+ and/or FISH/CISH-amplified).
3. Patients with any uncontrolled bleeding disorder including coagulation disorder or thrombocytopenia or prothrombotic disorder.
4. Patients with a personal history of autoimmune disease (including but not limited to multiple sclerosis, lupus, rheumatoid polyarthritis, inflammatory bowel diseases, Graves' disease and Hashimoto's disease).
5. Patients with a history of previous anaphylaxis or severe allergic reaction to vaccines or other known or unknown allergens.
6. Patients with previous splenectomy or radiation to the spleen.
7. Patients who have received a major organ graft (including bone-marrow transplantation).
8. Patients who require chronic oral treatment (defined as more than 14 days) with immunosuppressive agents including glucocorticosteroïds or other immune-modifying drugs. Use of topical and eye drops containing glucocorticosteroïds is acceptable, as well as inhaled corticosteroids.
9. Patients with previous or concomitant malignancies at other sites except effectively treated malignancy that has been in remission for >5 years and highly likely to have been cured. However patients with non-melanoma skin cancers or carcinoma in situ of the cervix can be included.
10. Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to unacceptable risk.
11. Patient with previous congestive heart failure or difficult-to-control hypertension and any uncontrolled vascular or cardiac disease.
12. Patient who has medically documented history of or active major depressive episode, bipolar disorders (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others).
13. Patient selects a response of "1,2 or 3" to question 9 on the PHQ-9 question regarding potential for suicidal thought or ideation (independent of the total score of PHQ-9)
14. Patient who has > CTCAE grade 3 anxiety.
15. Patients who have received (within 30 days before the inclusion) any investigational (biological or non-biological) or non-registered drug or non-registered vaccine other than the study vaccine, or who plan to receive such a drug during the study period.
16. Patients who have received any immunoglobulins and/or blood products within the 3 weeks prior to vaccine injection.
17. Patients who have received any commercial vaccine within one month before the first dose of study vaccine or are planned to receive any vaccine till 3 weeks after the 6th vaccine injection.
18. Patients who have out of range laboratory results as specified in the inclusion criteria.
19. Patients with a family history of congenital or hereditary immunodeficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
To assess the number of patient(s) presenting dose-limiting toxicities (DLTs) from the first vaccine injection in the first patient of the dose cohort till 3 weeks after the second vaccine injection of the last patient of the dose cohort. | 3 weeks after 2 study vaccine injections corresponding to visit number 5.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Leclerc, Study Chair — Institut Pasteur; Mario Campone, Principal Investigator — Institut de Cancérologie de l'Ouest (ICO)
Locations (5):
- France (5):
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'OUEST - Centre René Gauducheau, Nantes
  - Institut Curie, Paris
  - HEGP, Paris
  - Institut Gustave Roussy (IGR), Villejuif

REFERENCES:
- [Result] Rosenbaum P, Artaud C, Bay S, Ganneau C, Campone M, Delaloge S, Gourmelon C, Loirat D, Medioni J, Pein F, Sablin MP, Tredan O, Varga A, Leclerc C. The fully synthetic glycopeptide MAG-Tn3 therapeutic vaccine induces tumor-specific cytotoxic antibodies in breast cancer patients. Cancer Immunol Immunother. 2020 May;69(5):703-716. doi: 10.1007/s00262-020-02503-0. Epub 2020 Feb 7. PMID 32034426